CLINICAL TRIAL: NCT05305820
Title: The PANO Trial: Perioperative Exercise and Nutrition Optimisation Prehabilitation in Cancer Patients With Peritoneal Malignancy
Brief Title: Perioperative Exercise and Nutritional Optimisation Prehabilitation Before Surgery for Patients With Peritoneal Malignancy
Acronym: PANO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dublin City University (Other)
Collaborators: Mater Misericordiae University Hospital (Other); Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Aideen Scriney, Co-Investigator, Dublin City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: COALESE/2021/103; COALESE/2021/103 (Other Grant/Funding Number: Irish Research Council)
Record Dates: First submitted 2022-02-15; First posted 2022-03-31 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Peritoneal Malignancy; Ovarian Cancer; Rectum Cancer; Appendix Cancer; Colon Cancer
Keywords: Peritoneal Malignancy
MeSH Terms: conditions — Ovarian Neoplasms; Rectal Neoplasms; Appendiceal Neoplasms; Colonic Neoplasms | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Intervention Model Description: Parallel group randomised 1:1 controlled multi-centre trial
Masking Description: It will not be possible to be blinded to the to the allocation of participants due to their active involvement in the behavioural exercise and nutritional interventions during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Exercise: The exercise training program was designed to improve physical fitness prior to surgery and for a 6-week period after surgery once deemed fit.
  Nutrition: The nutritional arm consists of nutritional intervention tailored to the outcome of the nutritional screening.Participants will be asked to take part in a dietary food recall system called Foodbook24, and based on their dietary needs will be supported in nutritional optimisation.
  Interventions: Behavioral: Exercise; Behavioral: Nutrition
- Control (No Intervention): This group will receive standard oncological care and will receive no formal education of exercise or nutritional intervention.

INTERVENTIONS:
Behavioral: Exercise — Standard Exercise Program- Participants will be invited to take part in a structured home, supervised, or both, exercise program while undergoing treatment and for a six-week period when deemed fit post-surgery.
  Other Names: Tailored Exercise Prehabilitation Program
  Arms: Intervention
Behavioral: Nutrition — Participants will be screened for their nutritional health and tailored advice and education will be provided on an individualised basis. An online dietary recall tool will be used to track patients' dietary habits. This will occur from diagnosis until point of surgery and recommence for 6 weeks post-surgery once deemed physically fit.
  Other Names: Nutritional Optimisation
  Arms: Intervention

SUMMARY:
People who are diagnosed with cancer of the colon/rectum/appendix/ovaries that spreads into the lining of the tummy and some ovarian cancers or people with pseudomyxoma peritonei can often undergo intensive treatment including major surgery where chemotherapy is given whilst the person is having surgery - also known by doctors as surgery and hyperthermic intraperitoneal chemotherapy (HIPEC). Fitness for this surgery can improve if people undertake a prehabilitation programme at the time they get their diagnosis. To date, little research has focused on how exercise and nutrition support before surgery can help these patients during recovery. The aim of this study is to explore the use of exercise and nutritional support pre-treatment to enhance physical and psychological outcomes for patients.

DETAILED DESCRIPTION:
The comparator in this study will be standard oncological care. Control patients will receive the same care as standard without the addition of a formal exercise and nutrition support programme. The pre-treatment (prehabilitation) programme will commence following diagnosis and continue up to the point of surgery and recommence for six weeks following surgery when deemed clinically fit to participate. Assessments will occur at baseline, pre-surgery, post-surgery, and 6 weeks later and a follow up... Mixed methods will be employed with patients taking part in self-report assessments, physical assessments, and qualitative interviews. The primary aim of the study is to assess the feasibility of the intervention and cardiorespiratory fitness pre-surgery. The secondary aims include assessing the effect of the intervention on physical health, psychological wellbeing, health-related quality of life, self-efficacy, nutrition, and serology markers. Exploratory aims also include post-operative morbidity, health economics analysis and qualitative interview of patient experience.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* multidisciplinary team referral for CRS-HIPEC for colorectal/appendix/ovarian peritoneal disease or pseudomyxoma peritonei (+/- completed neoadjuvant cancer treatment)
* WHO performance status ≤2.

Exclusion Criteria:

* inability to provide informed consent,
* impaired cognitive function with a reduced ability to either understand advice /instructions from or communicate with the research team,
* declined surgery,
* surgery in less than 2 weeks
* pregnancy or breastfeeding,
* inability to participate in the exercise training (unable to perform the 6 Minute Walk Test)
* absolute contraindications to exercise testing, veganism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Adherence to the Intervention | 2-6 weeks pre surgery, 6 weeks post-surgery
  Prehabilitation fidelity in terms of the patient group adherence as measured by patient structured qualitative feedback and activity logs.
Feasibility of participant retention to the Intervention | 2-6 weeks pre-surgery, 6 weeks post-surgery
  Prehabilitation fidelity in terms of the patient group retention as measured by patient screening and retention logs and monitoring of recruitment rates.
Feasibility of intervention effectiveness | 2-6 weeks pre-surgery, 6 weeks post-surgery
  Prehabilitation fidelity in terms of intervention effectiveness as measured by qualitative patient feedback at two timepoints. Monitoring of patient activity logs. Engagement with online and in-person exercise and nutritional intervention resources.
Change in Cardiorespiratory Fitness | 2-6 weeks pre-surgery, 6 weeks post-surgery
  Cardiorespiratory fitness using the 6-Minute Walk Test (6MWT) assessed at the pre-surgery time point. The 6MWT is performed with participants walking up and down a 20 m course marked by cones for 6 min under instruction to cover as much ground as possible. The number of laps completed is recorded. A standard set of instructions is used as per the European Respiratory Society guidelines. The 6MWT is a validated assessment of cardiorespiratory function in clinical populations.

SECONDARY OUTCOMES:
Change in Strength - The Handgrip Test | 2-6 weeks pre-surgery, 6 weeks post-surgery
  This is measured using a hand dynamometer. The test will be conducted in a standing position with the upper arm tight against the participant's trunk and the forearm at a right angle to the upper arm. If this is not possible the participant may sit in an upright chair or use their free hand to rest the dynamometer on a table to support the arm. The gripping handle will be set to a comfortable width to ensure the patient can rest the middle piece of the four fingers on the handle. The participant will be instructed to squeeze the handle with maximum force for a few seconds. The value on the scale will be recorded. The participant will complete two trials on each hand. The highest score will be accepted.
Change in Strength - The Stand to Sit Test | 2-6 weeks pre-surgery, 6 weeks post-surgery
  Participants will sit on a chair (height 43-45 cm) with arms crossed on their, and legs flat on the floor, parallel to each other, and approximately shoulder width apart. Participants will stand up and sit down 10 times as quickly as possible. Participants must not bounce off the chair when moving from a seated position to standing position. They must fully extend their legs on each stand. The time taken to perform 10 repetitions will be timed using a stopwatch. Participants will perform two trials and the best trial will be recorded as their score.
Change in Activity - 3-day ActivPAL3 triaxial accelerometer | 2-6 weeks pre-surgery, 6 weeks post-surgery
  Participants will be instructed to wear the device on the midpoint of the anterior aspect of the right thigh and attach using a film adhesive frame dressing. They will continue to wear this for three days continuously. They cannot wear the ActivPAL3 triaxial accelerometer during water activity periods.
Change in Psychological Stress | 2-6 weeks pre-surgery, 6 weeks post-surgery
  NCCN Distress Thermometer: To detect distress (psychosocial stress) with all stages of cancer. This is measured using a visual analogue scale like a thermometer to indicate a range from 0 (not loaded) to 10 (extreme pressure). Additional 36 items in five problem areas - practical family, emotional, spiritual, physical, are rated for distress and a score of 5 or higher is considered significant stress.
Change in Psychological Stress- Impact of Events Scale | 2-6 weeks pre-surgery, 6 weeks post surgery
  This is a self-report measure of traumatic stress symptoms focused on intrusive thoughts and avoidant behaviours. Questions will be adapted to reflect the PM diagnosis specifically. Frequency of symptoms will be self-reported during the previous week using a 4 point scale from 0 (not at all) to 5 (often). Total scores range from 0 to 75 with higher scores indicative of greater cancer-related stress. Scores in the range of > 30 are reflective of clinically significant stress. Higher scores on an adapted IES are related to decreased immune function in breast cancer patients.
Change in Cognitive Reserve-Cognitive Reserve Index (CR-IQ) | 2-6 weeks pre-surgery, 6 weeks post surgery
  This questionnaire is a semi-structured interview with the patients that measures reserve in three parts: Education; Working-Activity, and Leisure time. Each sub-scale and total index score is correlated with age and expressed on a standardised scale.
Change in Cognition- FACT-Cog | 2-6 weeks pre-surgery, 6 weeks post surgery
  The Functional Assessment of Cancer Therapy- Cognition is a self-report 37 item questionnaire that assesses cancer related cognitive problems. Sub-scales include: Perceived cognitive impairments, impact of perceived cognitive impairments on QoL, Comments from others and perceived cognitive abilities.
Change in Self-Efficacy | 2-6 weeks pre-surgery, 6 weeks post surgery
  This is a 12 item Communication and Attitudinal Self-Efficacy scale for Cancer, and rates a patients' perceived ability to seek information, understand and engage in care, and maintain a positive attitude. Confidence level for each skill is rated on a 4 point scale with higher score indicative of higher self-efficacy.
Change in Health Related Quality of Life (HrQoL)-EQ-5D-5L (5L) | 2-6 weeks pre-surgery, 6 weeks post surgery
  This is a standardised and validated self-report measure describing health status. It is disease non-specific but applicable to cancer, with five dimensions (mobility, self-care, typical activities, pain, anxiety/depression) with three problem levels to rate (some to extremely problematic). The higher the index score, the higher the perceived health status.
Change in Health Related Quality of Life (HrQoL)- FACT-G | 2-6 weeks surgery, 6 weeks post surgery
  This is a version of the Functional Assessment of Cancer Therapy is a 28-item self-report survey that measures quality of life; it has 5 sub-scales measures physical well-being (PWB), functional wellbeing (FWB), social/family wellbeing (SFWB), emotional wellbeing (EWB) and satisfaction with care. Self-ratings of all 5 subscales for the present moment and the preceding week are captured, computing an overall total score. Good Cronbach's for all five have been reported, and the higher the core the better the QoL.
Change in Nutritional Status-The Malnutrition Screening Tool | 2-6 weeks pre-surgery, 6 weeks post surgery
  The Malnutrition Screening Tool (MST) is an easy to administer tool. It is based on recent appetite and weight loss and has been previously validated for use with oncology patients. The measure scores both "recent intake" and "recent weight loss". A total score of >2 indicates a risk of malnutrition.
Change in Nutritional Status- Glasgow Prognostic Score | 2-6 weeks pre-surgery, 6 weeks post surgery
  This measure of cancer prognosis is measured using serum markers CRP and Albumin. The score is used to measure the cancer prognosis. The score ranges from 0-2, with patients with a normal measure of CRP assigned a score of zero, and those with both elevated or reduced levels a score of 2.
Change in Dietary Intake - Foodbook24 | 2-6 weeks pre-surgery, 6 weeks post surgery
  Foodbook24 is a Web-based, dietary tool consisting of a 24-hour dietary recall and food frequency questionnaire. Patients will provide dietary recall information about what they have eaten in the past 24 hours.
Change in Nutritional Status- Blood Screening | 2-6 weeks pre-surgery, 6 weeks post surgery
  Bloods should be ordered by clinician for Iron (Fe) analysis (identify anaemia) and CT scans of patients should be analysed for the identification of incidence of sarcopenia.

OTHER OUTCOMES:
Post-operative Morbidity- Post-surgery Morbidity Score | Day 2 post
  This is an 18-item tool that addresses morbidity relevant to the post-surgical patient.
Post-operative Morbidity- The Clavien-Dindo classification | Day 15 post
  This is a classification of surgical complications with seven grades. The Comprehensive Complication Index (CCI) sums all post-operative complications with their respective severities on a scale of 0 (no burden) to 100 (fatality).
Post-Operative Morbidity- Comprehensive Complication Index | Day 15 post
  The Comprehensive Complication Index (CCI) sums all post-operative complications with their respective severities on a scale of 0 (no burden) to 100 (fatality).
Post-Operative Morbidity - Length of Hospital Stay | Day 1-15 post surgery
  Length of stay in hospital as a result of their operation.
Health Economic- Exploratory Analysis | 2-6 weeks pre surgery, 6 weeks post surgery
  An exploratory analysis will review healthcare resource use by individual participants and with locally determined unit cost calculate the healthcare cost related to the two interventions. The mean group difference in accumulated costs will be used in the cost-effectiveness analysis.
Serology Markers- Exploratory Analysis | 2-6 weeks pre-surgery, 6 weeks post surgery
  Biomarkers will be analysed on a sub-group (n=20) of recruited participants. Serological markers of inflammation using a multiplexed ELISA approach will be measured. The Luminex system can measure up to 45 serum cytokines and markers of inflammation, including the inflammatory cytokine IL-6, which has been associated with increased PS and PA. Inflammatory markers will be assessed at baseline, pre-surgery and post-surgery and 6 weeks post. Blood samples are taken routinely pre and post-surgery but for the purpose of the study the two additional timepoints of baseline/consent and 6 weeks post will also be taken. Using this dynamic approach, we will be able to correlate a patient's inflammatory response with their outcome during their prehabilitation and after surgery.
Qualitative Experience - Qualitative Patient Experience | 2-6 weeks pre surgery- 6 weeks post surgery
  Patients will also be asked whether they consent to take part in a short semi-structured phone interview with a member of the research team across two timepoints: pre surgery and 6 weeks post. The interviewer will ask the patients exploratory questions relating to four main topics: 1) Participants experiences and engagement with their care pathway (both control and intervention) 2) Perceptions of their emotional and physical preparation before surgery 3) Perceptions of their condition pre and post-surgery 4)Perceptions of physical and emotional symptoms pre and post-surgery.
Change in Smoking Status | 2-6 weeks pre surgery, 6 weeks post surgery
  Participants will be asked for their smoking status. If participants are active smokers who would like to cease smoking, they will be provided with the National Centre for Smoking Cessation and Training information support packages.

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Mulsow, Mr., Principal Investigator — Mater Misericordiae University Hospital; Lisa Loughney, Dr., Principal Investigator — Royal College of Surgeons, Ireland; Lorraine Boran, Dr., Principal Investigator — Dublin City University
Locations (3):
- Ireland (3):
  - Dublin City University, Dublin
  - Mater Misericordiae university hospital, Dublin
  - Royal College of Surgeons , Ireland, Dublin